CLINICAL TRIAL: NCT01061047
Title: Comparison of Ertapenem Distribution in the Muscle of Six Healthy Volunteers and Six Critically Ill Patients by Microdialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Other Study IDs: ERTAMUSCLE
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: patients infected with a bacteria sensible to ertapeneme

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ertapeneme

SUMMARY:
Ertapenem is an antibiotic that is highly bound to plasma protein (> 95%). The effects of this high protein binding on tissue distribution of antibiotics have been few evaluated yet.

In this study, two groups of subjects will be compared: 6 healthy volunteers and 6 critically ill patients (patients with infection due to an Ertapenem susceptible bacteria). Indeed, these 2 populations show changes in binding capacity of drugs to plasma proteins due to a decrease of protidaemia and of the affinity of drugs to transport proteins.

It seems therefore important to clarify the consequences of a modification in protein binding on distribution of antibiotics. That's why we have decided to characterize tissue distribution of ertapenem in healthy volunteers and critically ill patients by assessing: free and total concentrations in plasma and free concentrations in muscle by microdialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age: from 18 to 80 years
* Patients with infection due to ertapenem susceptible bacteria.

Exclusion Criteria:

* Patients who received ertapenem within 7 days prior to inclusion
* Known allergy to ertapenem or any excipients
* Neutropenia < 500/mm3
* Hemoglobin concentration < 9g/dl
* Renal failure (creatinin clearance < 30ml/min/1.73m²)
* Decompensated heart failure
* Patients receiving vasopressor (adrenalin, noradrenalin), > 0.5µg/kg/min
* Known hypersensitivity to Elma®
* Positive pregnancy test or currently lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital - 2 rue de la Milétrie - Réanimation chirugicale, Poitiers, France